CLINICAL TRIAL: NCT07377006
Title: Efforts to Enhance Germline Genetic Testing at Lyndon B. Johnson Hospital
Brief Title: Decision Support Tool to Enhance Germline Genetic Testing for Patients With Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-1272; NCI-2025-06571 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2025-1272 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2025-09-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Behavior Therapy; Specimen Handling; Genetic Counseling; Genetic Testing; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Qualitative interview) (Other): Patients complete a qualitative interview that informs the development of the decision support tool.
  Interventions: Other: Electronic Health Record Review; Other: Interview
- Group 2 (Draft decision support tool, cognitive interview) (Other): Patients view the draft of the decision support tool and complete cognitive interviews for the refinement of the decision support tool on study.
  Interventions: Behavioral: Behavioral Intervention; Other: Interview
- Group 3 (Decision tool) (Experimental): Patients view the decision support tool that provides culturally tailored information about genetic testing and the collection process. Patients may then provide a blood sample for standard of care genetic testing and may additionally meet with a genetics counselor for additional information prior to testing. Patients with a positive germline genetic mutation will discuss results with a genetics counselor.
  Interventions: Behavioral: Behavioral Intervention; Procedure: Biospecimen Collection; Other: Genetic Counseling; Other: Genetic Testing; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — View decision support tool
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Group 2 (Draft decision support tool, cognitive interview); Group 3 (Decision tool)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Group 3 (Decision tool)
Other: Electronic Health Record Review — Ancillary studies
  Arms: Group 1 (Qualitative interview)
Other: Genetic Counseling — Meet with genetic counselor
  Arms: Group 3 (Decision tool)
Other: Genetic Testing — Undergo standard of care genetic testing
  Other Names: Genetic Analysis; Genetic Examination; Genetic Test
  Arms: Group 3 (Decision tool)
Other: Interview — Complete qualitative interview
  Arms: Group 1 (Qualitative interview)
Other: Interview — Complete cognitive interview
  Arms: Group 2 (Draft decision support tool, cognitive interview)
Other: Survey Administration — Ancillary studies
  Arms: Group 3 (Decision tool)

SUMMARY:
This clinical trial identifies factors associated with completing genetic testing, aids in the development of a decision support tool, and tests how well the decision support tool works to enhance germline genetic testing in patients with prostate cancer. Germline genetic testing is a guideline-recommended standard of care for many patients with prostate cancer. Completing genetic testing can enable the use of targeted therapies, offers access to novel clinical trials, provides valuable information, and can help identify at risk family members. The decision support tool may educate patients and assist in the decision to engage with germline genetic testing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify patient, provider, and health system factors contributing to the completion of recommended germline testing for men with prostate cancer.

II. Develop a decision support tool for patients tailored to the cultural and socioeconomic context of the local community.

III. Conduct a pilot intervention trial to evaluate a point-of-care decision support tool in a public safety net hospital in Harris County, Texas.

SECONDARY OBJECTIVES:

I. Assess the feasibility of point-of-care decision support tool in a public safety net hospital in Harris County, Texas.

II. Assess the change in completion of germline genetic testing with utilization of the decision support tool.

OUTLINE: At each stage of the proposed research, patients are recruited to 1 of 3 groups. Groups 1 and 2 are observational and group 3 is a pilot interventional trial.

GROUP 1: Patients complete a qualitative interview that informs the development of the decision support tool.

GROUP 2: Patients view the draft of the decision support tool and complete cognitive interviews for the refinement of the decision support tool on study.

GROUP 3: Patients view the decision support tool that provides culturally tailored information about genetic testing and the collection process. Patients may then provide a blood sample for standard of care genetic testing and may additionally meet with a genetics counselor for additional information prior to testing. Patients with a positive germline genetic mutation will discuss results with a genetics counselor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed prostate cancer patients receiving care at Lyndon B. Johnson (LBJ) Hospital
* Were recommended for germline genetic testing by their oncology provider
* Can provide informed consent
* Can communicate in English or Spanish

Exclusion Criteria:

* Prostate cancer patients receiving care at LBJ who are unable to participate due to a serious psychological or cognitive condition

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Debanjan Pain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States